CLINICAL TRIAL: NCT02042443
Title: Randomized Phase II Trial of Single Agent MEK Inhibitor Trametinib (GSK1120212) Vs 5-Fluorouracil or Capecitabine in Refractory Advanced Biliary Cancer
Brief Title: Trametinib or Combination Chemotherapy in Treating Patients With Refractory or Advanced Biliary or Gallbladder Cancer or That Cannot Be Removed by Surgery
Acronym: S1310
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-02485; NCI-2013-02485 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1310; SWOG-S1310; S1310 (Other: SWOG); S1310 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: Adult Cholangiocarcinoma; Advanced Adult Hepatocellular Carcinoma; BCLC Stage C Adult Hepatocellular Carcinoma; BCLC Stage D Adult Hepatocellular Carcinoma; Hilar Cholangiocarcinoma; Localized Non-Resectable Adult Liver Carcinoma; Recurrent Adult Liver Carcinoma; Recurrent Childhood Liver Cancer; Recurrent Extrahepatic Bile Duct Carcinoma; Recurrent Gallbladder Carcinoma; Stage II Gallbladder Cancer; Stage III Childhood Hepatocellular Carcinoma; Stage IIIA Gallbladder Cancer; Stage IIIB Gallbladder Cancer; Stage IV Childhood Hepatocellular Carcinoma; Stage IV Distal Bile Duct Cancer; Stage IVA Gallbladder Cancer; Stage IVB Gallbladder Cancer; Unresectable Extrahepatic Bile Duct Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Klatskin Tumor; Carcinoma, Hepatocellular; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Capecitabine; Fluorouracil; dehydroftorafur; Leucovorin; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trametinib (Experimental): Patients receive trametinib PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Trametinib
- Chemotherapy (Experimental): Patients receive either A) leucovorin calcium IV over 2 hours and fluorouracil IV continuously over 46-48 hours on days 1 and 15 (courses repeat every 28 days); or B) capecitabine PO BID on days 1-14 (courses repeat every 21 days). Patients treated until disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
  Arms: Chemotherapy
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Chemotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Chemotherapy
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist
  Arms: Trametinib

SUMMARY:
This randomized phase II trial studies how well trametinib or combination chemotherapy works in treating patients with refractory or advanced biliary or gallbladder cancer or that cannot be removed by surgery. Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fluorouracil, leucovorin calcium, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving trametinib is more effective than combination chemotherapy in treating patients with biliary or gallbladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess overall survival (OS) in patients with refractory advanced biliary cancer randomized to Arm 1: trametinib compared to those randomized to Arm 2: chemotherapy (either 5-fluorouracil [fluorouracil] and leucovorin [leucovorin calcium] or capecitabine).

SECONDARY OBJECTIVES:

I. To determine the frequency and severity of adverse events of trametinib in this patient population.

II. To assess response rate (RR) and progression-free survival (PFS) in patients randomized to Arm 1: trametinib and patients randomized to Arm 2: chemotherapy (fluorouracil [5-FU] or capecitabine in this patient population).

TERTIARY OBJECTIVES:

I. To determine if a 16-gene expression signature is predictive of mitogen-activated protein kinase kinase (MEK) efficacy as evidenced by improved RR, PFS, and OS.

II. To evaluate the effects of trametinib on the inflammatory cytokine and explore potential associations with response rate and survival.

III. To estimate lean soft tissue and fat mass weight gain as a result of treatment with trametinib vs. capecitabine in patients with advanced refractory biliary cancer.

IV. To bank tissue samples for other future correlative studies including next generation sequencing and whole genome methylation assays. NOTE: These potential future correlative studies will not be performed until an amended protocol with relevant detailed information including specific arms and assays is approved by Cancer Therapy Evaluation Program (CTEP).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive trametinib orally (PO) once daily (QD) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive 1 of 2 treatment regimens at the discretion of the investigator.

ARM IIA: Patients receive leucovorin calcium intravenously (IV) over 2 hours and fluorouracil IV continuously over 46-48 hours on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM IIB: Patients receive capecitabine PO twice daily (BID) on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* DISEASE RELATED CRITERIA
* Patients must have histologically or cytologically documented carcinoma primary to the intra- or extra-hepatic biliary system or gall bladder with clinical and/or radiologic evidence of unresectable, locally advanced or metastatic disease; patients with ampullary carcinoma are not eligible
* Patients must have measurable disease; computed tomography (CT) scans or magnetic resonance imaging (MRI)s used to assess measurable disease must have been completed within 28 days prior to registration; CT scans or MRIs used to assess non-measurable disease must have been completed within 42 days prior to registration; all disease must be assessed and documented on the Baseline Tumor Assessment Form (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)
* PRIOR/CONCURRENT THERAPY CRITERIA
* Patients must have completed any prior chemotherapy at least 21 days prior to registration and have recovered from any of the effects AND

  * Patients must have experienced progression to no more than 1 prior regimen of systemic chemotherapy for advanced biliary cancer OR
  * Patients who received adjuvant chemotherapy and had evidence of disease recurrence within 6 months of completion of the adjuvant treatment are also eligible; if patient received adjuvant treatment and had disease recurrence after 6 months, patients will only be eligible after failing one regimen of systemic chemotherapy used to treat the (unresectable or metastatic) disease recurrence
* Patients must not have been treated with prior MEK inhibitors; prior 5-FU or capecitabine treatment is allowed only if given as a radiosensitizer concurrently with radiation therapy at least 12 weeks prior to registration or if given as part of any adjuvant therapy regimen >= 12 months prior to study enrollment
* Patients must have no plans to receive concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy or any other type of therapy (including herbal or natural supplements) for treatment of cancer while on this treatment protocol
* For patients who have received prior cryotherapy, radiation therapy, radiofrequency ablation, therasphere, ethanol injection, transarterial chemoembolization (TACE) or photodynamic therapy, the following criteria must be met:

  * 28 days have elapsed since that therapy (lesions that have not been treated with local therapy must be present and measureable)
* CLINICAL/LABORATORY CRITERIA
* Patients must have a Zubrod performance status of 0-1
* Absolute neutrophil count (ANC) > 1000/mcL
* Platelets > 100000/mcL
* Total bilirubin =< 2.0 x the institutional upper limit of normal limits (IULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both =< 3 x IULN; if liver metastases are present, AST and ALT must be =< 5 x IULN
* If the patient has had decompression of the biliary tree within the last 14 days, stability of the bilirubin level needs to be confirmed with two measurements that are within 5 to 7 days of each other; (the second measurement must be obtained within 7 days prior to registration;) both the first and second measurement must be =< 2.0 x IULN; stability is defined as the second measurement being no more than one point higher than the first
* Patients must have adequate kidney function as evidenced by at least ONE of the following:

  * Serum creatinine =< 1.5 x IULN within 28 days prior to registration
  * Calculated creatinine clearance >= 50 ml/min for patients with creatinine level of 1.0-1.5 x IULN; the serum creatinine value used in the calculation must have been obtained within 28 days prior to registration
* Patients with known history or current evidence of retinal vein occlusion (RVO) or retinal pigment epithelial detachment (RPED) are not eligible:

  * History of RVO or RPED, or predisposing factors to RVO or RPED (e.g. such as uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes)
  * Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or RPED such as:

    * Evidence of new optic disc cupping
    * Evidence of new visual field defects
    * Intraocular pressure > 21 mmHg
  * NOTE: ophthalmic exam is required for all patients; this exam should not be performed until or unless it is very clear the patient is otherwise eligible for registration; this exam should not be performed until or unless it is very clear the patient is otherwise eligible for registration
* Patients must have echocardiogram and left ventricular ejection fraction (LVEF) >= institutional lower limit of normal (LLN) within 28 days prior to registration; this exam should not be performed until or unless it is very clear the patient is otherwise eligible for registration
* Patients must not have uncontrolled or clinically significant cardiovascular disease including: myocardial infarction within past 6 months; uncontrolled angina within past 6 months; class II-IV New York Heart Association (NYHA) congestive heart failure; grade 3 cardiac valve dysfunction; cardiac arrhythmia not controlled by medication; history of stroke or transient ischemic attack within 6 months; history of arterial thrombotic event (ATE) of any type in the past 6 months; treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled with anti-hypertensive therapy; known intra-cardiac defibrillators; known cardiac metastases
* Patients must have an electrocardiogram (ECG) within 28 days prior to registration; patients must have corrected QT interval (QTc) =< 500 msec; this exam should not be performed until or unless it is very clear the patient is otherwise eligible for registration
* Must be able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Must not have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib, or excipients or to dimethyl sulfoxide (DMSO) or other agents used in study
* Must not have active hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (patients with chronic or cleared HBV and HCV infection are eligible)
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method while on study and for 4 months after discontinuation of study drug; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* SPECIMEN SUBMISSION CRITERIA
* Patients must submit paraffin-embedded tissue and blood for banking within 28 days after registration; paraffin-embedded tissue from prior surgical resection or from a diagnostic biopsy is acceptable
* REGULATORY CRITERIA
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-02; Primary Completion 2017-01 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, Principal Investigator — SWOG Cancer Research Network
Locations (295):
- United States (295):
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Hospital, Fontana, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente, Woodland Hills, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Medical Oncology and Hematology Group PC-Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Charlotte Hungerford Hospital Center for Cancer Care, Torrington, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - University of Florida, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Reid Health, Richmond, Indiana
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - The University of Kansas Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology - Fort Apache, Las Vegas, Nevada
  - Cancer and Blood Specialists-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - 21st Century Oncology - Vegas Tenaya, Las Vegas, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Asheville Hematology-Oncology Associates, Asheville, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Roper Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates-Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Charleston Hematology Oncology Associates PA-St. Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Kingsport, Kingsport, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - The Methodist Hospital System, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy: Patients receive either A) leucovorin calcium IV over 2 hours and fluorouracil IV continuously over 46-48 hours on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity or B) capecitabine PO BID on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Trametinib | Chemotherapy
Started | 27 | 26
Eligible and Analyzable | 24 | 20
Completed | 0 | 0
Not Completed | 27 | 26
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Progression | 21 | 17
Not completed — not protocol specified | 1 | 1
Not completed — Not eligible/not analyzable | 3 | 6

BASELINE CHARACTERISTICS:
Population: All eligible and analyzable patients are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trametinib | Chemotherapy | Total
Number analyzed (Participants) | 24 | 20 | 44
Age, Continuous [Median (Full Range); unit: years] | 63 [40 to 78] | 61 [41 to 81] | 62 [40 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 11 | 29
  Male | 6 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Planned Chemotherapy [Count of Participants; unit: Participants]
  5FU/LV | 7 | 6 | 13
  Capecitabine | 17 | 14 | 31
Site of Disease [Count of Participants; unit: Participants]
  Cholangiocarcinoma | 19 | 15 | 34
  Gall bladder | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Up to 2 years from registration
Population: Eligible and analyzable patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 24 | 20
months | 4.3 [3.1 to 5.1] | 7.9 [3.2 to 14.6]
Statistical Analysis 1: Comparison: Trametinib vs Chemotherapy; Test type: Superiority; p = 0.05, Log Rank; Hazard Ratio (HR) = 2.02, 95% CI 2-sided [1.01 to 4.03]

2. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse event reporting followed the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 4.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 2 years
Population: Eligible patients who received any treatment and were assessed for adverse events are included in this summary. One patient was hospitalized prior to receiving protocol treatment and was not assessed for adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 23 | 20
Participants
  Alanine aminotransferase increased | 1 | 0
  Anemia | 1 | 0
  Ascites | 1 | 0
  Aspartate aminotransferase increased | 1 | 0
  Blood bilirubin increased | 1 | 0
  Colitis | 0 | 1
  Fatigue | 0 | 1
  Gastric ulcer | 1 | 0
  Gastritis | 1 | 0
  Gastrointestinal disorders - Other, specify | 1 | 0
  Generalized muscle weakness | 0 | 1
  Hepatobiliary disorders - Other, specify | 1 | 0
  Hyponatremia | 1 | 1
  Infections and infestations - Other, specify | 0 | 1
  Mucositis oral | 0 | 1
  Neutrophil count decreased | 0 | 1
  Pain in extremity | 0 | 1
  Palmar-plantar erythrodysesthesia syndrome | 0 | 1
  Sepsis | 1 | 0
  Thromboembolic event | 1 | 0
  Urinary tract infection | 1 | 0
  Vomiting | 1 | 0

3. Secondary Outcome: Objective Response Rate
Description: Confirmed response (CR) is two or more objective statuses of CR a minimum of four weeks apart documented before progression or symptomatic deterioration. Partial response (PR) is two or more objective statuses of PR or better a minimum of four weeks apart documented before progression or symptomatic deterioration. Unconfirmed CR is one objective status of CR documented before progression or symptomatic deterioration but not qualifying as CR or PR. Unconfirmed PR is one objective status of PR documented before progression or symptomatic deterioration but not qualifying as CR, PR or unconfirmed CR.
Time Frame: Up to 2 years from registration
Population: All eligible and analyzable patients with measurable disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 24 | 20
Participants
  Partial Response | 0 | 2
  Unconfirmed Partial Response | 2 | 0
  Stable/No Response | 2 | 9
  Increasing Disease | 19 | 8
  Symptomatic Deterioration | 1 | 1

4. Secondary Outcome: Progression-free Survival
Description: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression free are censored at date of last contact.
Time Frame: Up to 2 years from registration
Population: Eligible and analyzable patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 24 | 20
months | 1.3 [1.2 to 1.5] | 2.8 [1.4 to 6.9]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Eligible patients who received any treatment and were assessed for adverse events are included in the adverse event summaries. One patient was hospitalized prior to receiving protocol treatment and was not assessed for adverse events.
Arm/Group | Trametinib | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 13/23 | 1/20
Other Adverse Events (participants affected / at risk) | 21/23 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trametinib (N=23) | Chemotherapy (N=20)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 2 | 0
Hepatobiliary disorders-Other (Hepatobiliary disorders) | 1 | 0
Infections and infestations-Other (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trametinib (N=23) | Chemotherapy (N=20)
Anemia (Blood and lymphatic system disorders) | 8 | 8
Ear and labyrinth disorders-Other (Ear and labyrinth disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Dry eye (Eye disorders) | 3 | 2
Watering eyes (Eye disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 4
Ascites (Gastrointestinal disorders) | 1 | 1
Bloating (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 6
Diarrhea (Gastrointestinal disorders) | 4 | 7
Dry mouth (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 7 | 8
Vomiting (Gastrointestinal disorders) | 7 | 5
Chills (General disorders) | 4 | 1
Edema limbs (General disorders) | 4 | 4
Fatigue (General disorders) | 11 | 11
Fever (General disorders) | 4 | 4
Irritability (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 6 | 6
Infections and infestations-Other (Infections and infestations) | 1 | 2
Papulopustular rash (Infections and infestations) | 2 | 1
Paronychia (Infections and infestations) | 0 | 1
Rhinitis infective (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 3
Alanine aminotransferase increased (Investigations) | 6 | 0
Alkaline phosphatase increased (Investigations) | 6 | 3
Aspartate aminotransferase increased (Investigations) | 8 | 5
Blood bilirubin increased (Investigations) | 3 | 5
Creatinine increased (Investigations) | 1 | 4
Investigations-Other (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 3
Neutrophil count decreased (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 6 | 6
Weight loss (Investigations) | 0 | 2
White blood cell decreased (Investigations) | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 5 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 3
Hyponatremia (Metabolism and nutrition disorders) | 2 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Dizziness (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 3 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3
Presyncope (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Confusion (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 1
Urine discoloration (Renal and urinary disorders) | 2 | 2
Breast pain (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 5
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 14 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 6 | 3
Hypotension (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less